CLINICAL TRIAL: NCT05229328
Title: Study on the Establishment of a System for Early Warning and Prognostic Evaluation
Brief Title: Study on the Establishment of a System for Early Warning and Prognostic Evaluation of Patients With Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20212172
Record Dates: First submitted 2021-11-14; First posted 2022-02-08 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-11

CONDITIONS: Sepsis; Prognosis; Liver Injury; Kidney Injury; Early Waking
MeSH Terms: conditions — Sepsis; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, PBMC, plasma exosome miRNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Healthy volunteers
  Interventions: Diagnostic Test: Peripheral blood test
- Patients within the acute phase of disease: Patients within 24 hours after onset
  Interventions: Diagnostic Test: Peripheral blood test
- Recovery phase of disease: Inflammation was controlled, shock was corrected, and the patient remained fever free for 3 consecutive days.
  Interventions: Diagnostic Test: Peripheral blood test

INTERVENTIONS:
Diagnostic Test: Peripheral blood test — Collect peripheral blood to separate and extract plasma, PBMC, and plasma exosomal miRNA, and sequence to find indicators related to disease deterioration and prognosis

SUMMARY:
Sepsis is a clinical syndrome with high morbidity and high fatality rate in emergency department. Patients with acute liver or kidney injury are more likely to develop Multiple Organ Dysfunction Syndrome(MODS) secondary to the non-hepatic injury group, and the prognosis deteriorates significantly. At present, there is no unified diagnostic criteria for acute liver injury associated with sepsis, and the commonly used prognostic evaluation system is rarely included in liver injury indicators, which is not good for practicality.

DETAILED DESCRIPTION:
The project intends to collect the peripheral blood of the normal population, 24 hours after the onset of sepsis and patients in the recovery period. We will separate and extract plasma, Peripheral Blood Mononuclear Cell(PBMC), and plasma exosomal miRNA, and sequence to find indicators related to disease deterioration and prognosis. And then, we will construct and verify the early warning and prognosis evaluation system.

On this basis, the researcher explore cellular and molecular mediated pathological mechanisms of sepsis, and then clarify the treatment target of sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. The patient who voluntarily signs an informed consent form;
2. Adult patients who meet the criteria for sepsis, who is registration to the hospital within 24 hours of onset;
3. SEPSIS is defined as the sequential organ failure assessment (SOFA) score ≥ 2 within 24 hours after admission, accompanied by at least one site of infection;
4. Patients with septic shock can be identified with a clinical construct of sepsis with persisting hypotension requiring vasopressors to maintain mean arterial pressure(MAP) 65 mm Hg and having a serum lactate level >2 mmol/L (18 mg/dL) despite adequate volume resuscitation.

Exclusion Criteria:

1. Age <18 years old or >90 years old;
2. Patients with advanced tumors, Pregnancy or lactation;
3. Patients who missed out during treatment and whose data are incomplete.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Healthy Volunteers;
  2. Adult patients who meet the criteria for sepsis, defined as life-threatening organ dysfunction caused by a dysregulated host response to infection.
  3. Septic shock is a subset of sepsis in which underlying circulatory and cellular/metabolic abnormalities are profound enough to substantially increase mortality.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Surviving or Died Participants with sepsis | Day 30
  Prognosis
Rate of Surviving or Died Participants with sepsis | Day 90
  Prognosis

SECONDARY OUTCOMES:
Sepsis-associated liver injury | Day 0
  Concentration of Alanine aminotransferase(ALT) >80 U/L or Glutamine oxaloacetic transaminase (GOT,AST) >80 U/L, Concentration of total bilirubin(TBIL)>2mg/dl（34μmol/l）
Sepsis-associated kidney injury | Day 0
  Concentration of Creatinine(Cr)>2 mg/dl or Urine output < 500ml/Day

CONTACTS AND LOCATIONS:
Overall Officials: Yanyan Jia, Study Chair — The First Affillated Hospital,the Air Force Medical University
Locations (1):
- The First Affillated Hospital,the Air Force Medical University, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: No